CLINICAL TRIAL: NCT04945200
Title: Neoadjuvant Immune Checkpoint Inhibitor Combined With Chemotherapy in Non-small Cell Lung Cancer: Clinical Response and Biomarkers Analysis
Brief Title: Neoadjuvant Immune Checkpoint Inhibitor Combined With Chemotherapy in Non-small Cell Lung Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-1003
Record Dates: First submitted 2021-06-17; First posted 2021-06-30 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-03

CONDITIONS: Non-small Cell Lung Cancer
Keywords: non-small cell lung cancer, neoadjuvant, biomarker
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The primary object of this study is to determine tumor major pathological response (MPR) rate and pathologic complete response (pCR) rate in stage IB-IIIA non-small cell lung cancer who subjected to neoadjuvant immune checkpoint inhibitor combined with chemotherapy and molecular biomarkers related to the clinical response.

ELIGIBILITY:
Inclusion Criteria:

1.Able to understand the nature of this trial and provide written informed consent.

2.18 years ≤ age ≤ 80 years

3.Histologically documented non-small cell lung cancer

4.NSCLC with resection option for potential cure.This may include clinical stage IB, II and IIIA.

5.Subjected to neoadjuvant immune checkpoint inhibitor combined with chemotherapy according to disease evaluation.

6.Measurable disease by RECIST v1.1

7.Tumor tissue sample and/or alveolar lavage fluid must be available for biomarker evaluation before operation.

Exclusion Criteria:

1. Subjects are excluded if they are enrolled in any other interventional studies.
2. Administration of chemotherapy, device therapy or any other cancer therapy in 4 weeks before the study drug administration.
3. Subjects are excluded if they have an active, known or suspected autoimmune disease requiring systemic treatment (e.g.corticosteroids or other immunosuppressive medications) in 2 years before the study drug administration. substitution therapy ( e.g. thyroxine, insulin) are permitted.
4. Subjects with active concurrent malignancies are excluded i.e. cancers other than NSCLC.
5. History of allergy to study drug components
6. Any other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or may interfere with the interpretation of study results.
7. Any other conditions that, in the Investigator's opinion, unfit to attend this study.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: stage IB-IIIA NSCLC
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
molecular biomarkers related to clinical response | change from baseline to postoperation, an average of 1 week
  molecular biomarkers related to tumor major pathological response (MPR) and pathologic complete response (pCR) in stage IB-IIIA non-small cell lung cancer who subjected to neoadjuvant immune checkpoint inhibitor combined with chemotherapy

CONTACTS AND LOCATIONS:
Locations (1):
- 2nd Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China